CLINICAL TRIAL: NCT01637090
Title: PHASE II TRIAL OF THE mTOR INHIBITOR EVEROLIMUS IN RELAPSED OR REFRACTORY CUTANEOUS T-CELL LYMPHOMA (CTCL)
Brief Title: Everolimus in Treating Cutaneous T-cell Lymphoma
Acronym: CTCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Adam Lerner (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Adam Lerner, Principal Investigator, Boston Medical Center
Organization: Boston Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-30213
Record Dates: First submitted 2012-04-02; First posted 2012-07-10 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cutaneous T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- all patients on study (Experimental): This will be a prospective, phase II non-randomized, open label study of single agent everolimus for the treatment of CTCL recurrent or refractory to at least one previous treatment other than topical medication. The purpose will be evaluation of safety and anti-tumor response as evaluated by serial skin examinations and assessment of tumor burden in tissue and blood.
  This study will be conducted in 2 stages. During stage 1 we will enroll a maximum of 11 subjects to evaluate response rate and will only continue to stage 2, if we observe two or more responses. During stage 2, we will expand the study to an overall N of 28 patients.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — The study drug everolimus will be self-administered (by the patients themselves). The investigator will instruct the patient to take the study drug exactly as specified in the protocol. Everolimus should be administered orally once daily, preferably in the morning, at the same time every day with our without food. Everolimus tablets should be swallowed whole with a glass of water. The tablets must not be chewed or crushed.
  Everolimus will be administered orally as once daily dose of 10 mg continuously from study day 1 until progression of disease or unacceptable toxicity.
  If vomiting occurs, no attempt should be made to replace the vomited dose. All dosages prescribed and dispensed to the patient and all dose changes during the study must be recorded.
  Other Names: Afinitor

SUMMARY:
CTCL is a rare form of lymphoma of the skin. While early stages are usually confined to the skin, later stages may spread to blood, lymph nodes and other organs. At this point, patients usually require systemic chemo. This study will investigate the effect of everolimus as treatment for recurrent or refractory CTCL. Participation in this study will last as long as the study doctor believes disease has not gotten worse, and patients continue to tolerate the study medication for a maximum of 1 year. Once off the treatment, patients will be followed for two years.

DETAILED DESCRIPTION:
Cutaneous T-cell lymphoma is a rare form of lymphoma of the skin. While early stages are usually confined to the skin, later stages may spread to blood, lymph nodes and other organs. At this point, patients usually require systemic chemotherapy. This study will investigate the effect of everolimus as a treatment for patients diagnosed with CTCL that has either not responded to previous treatments or has recurred despite previous treatments. Everolimus is the common name for the commercial drug Afinitor® (Novartis). It is approved by the U.S. Food and Drug Administration (FDA) for use in kidney and brain cancer. In several different forms of lymphomas, everolimus is used as an investigational drug, which means it has not been approved by the FDA for this group of diseases.

Everolimus blocks a protein (mTOR) that helps cells and tumors to grow. Earlier studies have indicated that the drug everolimus may work against lymphomas including cutaneous T-cell lymphomas. Participation in this study will last as long as the study doctor believes disease has not gotten worse, and patients continue to tolerate the study medication for a maximum of 1 year. Once off the treatment, patients will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and histologically confirmed diagnosis of CTCL (at least stage IB for mycosis fungoides and Sézary syndrome, and T2 and/or refractory to at least one prior treatment for CTCL other than mycosis fungoides/Sézary syndrome)
* Relapsed or refractory disease after at least one standard systemic treatment including extracorporeal photopheresis (ECP), oral bexarotene, interferon, HDAC inhibitors
* ≥18 years old
* WHO performance status ≤ 2
* Life expectancy ≥ 6 months
* ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Serum bilirubin ≤ 1.5 x ULN
* ALT and AST ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
* INR ≤1.5 (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of randomization)
* Serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L
* Fasting triglycerides ≤ 2.5 x ULN.

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of stating study drug
* Treatment with any investigational drug within the past 4 weeks
* Patients, who have had major surgery or significant traumatic injury within 4 weeks of starting study drug, patients who have not recovered from the side effects of any major surgery, or patients that may require major surgery during the study
* Patients receiving chronic, systemic treatment with corticosteroids or any immunosuppressive agent other than topical or inhaled corticosteroids
* Patients receiving immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Symptomatic congestive heart failure of New York heart Association Class III or IV
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
* uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN (Note: Optimal glycemic control should be achieved before starting trial therapy.)
* active (acute or chronic) or uncontrolled severe infections
* liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes.
* Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients who have received prior treatment with an mTOR inhibitor
* Patients with a known hypersensitivity to everolimus or other rapamycins or to its excipient
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lerner, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was actively recruiting from within the investigator's own praceice from June 2012 through May 2015 in the hematology/oncology multidisciplinary clinic.
Groups:
- All Patients on Study: Prospective, phase II non-randomized, open label study of single agent everolimus for the treatment of CTCL recurrent or refractory to at least one previous treatment other than topical medication. The purpose will be evaluation of safety and anti-tumor response as evaluated by serial skin examinations and assessment of tumor burden in tissue and blood.
  This study will be conducted in 2 stages. During stage 1 we will enroll a maximum of 11 subjects to evaluate response rate and will only continue to stage 2, if we observe two or more responses. During stage 2, we will expand the study to an overall N of 28 patients.
  Everolimus will be administered orally as once daily dose of 10 mg continuously from study day 1 until progression of disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | All Patients on Study
Started | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Patients on Study
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — greater than or equal to 18 years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 1
    >=65 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Treatment
Description: Determine the efficacy of everolimus in the treatment of CTCL as overall response rate (ORR)
Time Frame: 12 months after beginning treatment
Population: Study was pre-maturely terminated. No data were collected for the Outcome Measure
Arm/Group | All Patients on Study
Number analyzed (Participants) | 0
Value | 0

2. Secondary Outcome: Time to Response
Description: Determine time to response (TTR)/duration of objective response (DOR)
Time Frame: three months
Population: Study was pre-maturely terminated. No data were collected for the Outcome Measure
Arm/Group | All Patients on Study
Number analyzed (Participants) | 0
Value | 0

3. Secondary Outcome: Progression-free Survival
Description: Determine progression-free survival of CTCL patients treated with everolimus
Time Frame: two years after discontinuing study treatment
Population: Study was pre-maturely terminated. No data were collected for the Outcome Measure
Arm/Group | All Patients on Study
Number analyzed (Participants) | 0
Value | 0

4. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Determine the adverse event profile and tolerability of everolimus in patients with CTCL
Time Frame: Up to one year
Measure: Number; unit: participants
Arm/Group | All Patients on Study
Number analyzed (Participants) | 3
participants | 3

5. Secondary Outcome: Effect of mTOR on Tumors
Description: Determine mTOR (mammilian target of rapamycin) pathway activation and number of regulatory T cells (Tregs) in pre-treated tumor tissue and evaluate changes following treatment
Time Frame: one year
Population: Study was pre-maturely terminated. No data were collected for the Outcome Measure
Arm/Group | All Patients on Study
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Time Frame: Adverse event reporting was to be collected for up to one year.
Arm/Group | All Patients on Study
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients on Study (N=3)
fatigue (General disorders) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1
skin infection (Infections and infestations) | 1 (1) — cellulitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes